CLINICAL TRIAL: NCT05451381
Title: Vasopressor Requirements During Dexmedetomidine Sedation vs Propofol vs Their Combination (Dexmedetomidine and Propofol) Sedation in Patients After Cardiac Surgery
Brief Title: Vasopressor Requirements Depends on Sedation Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anesthesia Research Group UA (Other)
Responsible Party: Principal Investigator, Plechysta Yelyzaveta, chief of the anesthesia department, Anesthesia Research Group UA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0120U100657
Record Dates: First submitted 2022-06-21; First posted 2022-07-11 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Sedative Adverse Reaction; Sedation Complication; Hemodynamic Instability; Agitation on Recovery From Sedation; Respiratory Complication
MeSH Terms: interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol group (Experimental): Patient sedation after cardiac surgery at the intensive care unit.
  Sedation group (PR):
  continuous infusion of propofol using a syringe pump at the dose of 1-1.5 mg / kg / h
  Interventions: Drug: Propofol
- Dexmedetomidine group (Experimental): Patient sedation after cardiac surgery at the intensive care unit.
  Sedation group Dexmedetomidine (DEX):
  continuous infusion of Dexmedetomidine using a syringe pump at the dose of 0.5-1.0 mcg/ kg / h
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine and propofol group (Experimental): Patient sedation after cardiac surgery at the intensive care unit.
  Sedation group DEX+PR:
  continuous infusion of propofol using a syringe pump at the dose of 0.5-1.5 mg / kg / h and dexmedetomidine 0.2-0.7 mcg\kg\h
  Interventions: Drug: Dexmedetomidine and Propofol

INTERVENTIONS:
Drug: Propofol — sedation after cardiac surgery
  Other Names: PR
  Arms: Propofol group
Drug: Dexmedetomidine — sedation after cardiac surgery
  Other Names: DEX
  Arms: Dexmedetomidine group
Drug: Dexmedetomidine and Propofol — sedation after cardiac surgery
  Other Names: DEX+PR
  Arms: Dexmedetomidine and propofol group

SUMMARY:
Most of the patients after cardiac surgery need sedation in the iCU. Sedation strategy could impact the incidence of vasopressor use.

DETAILED DESCRIPTION:
Sedating a patient is a complex process, especially after heart surgery. Sedation has a negative hemodynamic effect. This leads to a decrease in blood pressure and increases the frequency and dose of vasopressors used. The choice of drug for sedation may have an impact on reducing the frequency of use of vasopressor therapy. The goal of the research is compare three strategies: propofol ( sedative agent), dexmedetomidine ( selective α2-adrenergic receptor (α2-AR) agonist that is associated with sedative effect) and their combination for sedation after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Multi vascular lesions of the coronary arteries according to coronary angiography;
* Heart valve damage was confirmed by heart ultrasound, which is subject to surgical correction (aortic stenosis of III degree with a gradient on the aortic valve of more than 42 mmHg, aortic insufficiency III, mitral valve stenosis II-III, mitral regurgitation II-III)
* Age of patients from 18-80 years;
* Patient consent to participate in the study;
* Women who have a negative pregnancy test and use effective contraception throughout the study and for 3 weeks after its completion, or women who are unable to have children (women who have undergone a hysterectomy (removal of the uterus) or tubal ligation, women with a clinical diagnosis of infertility) or are menopausal for more than 1 year (absence of menstruation for at least 12 months). Adequate methods of contraception include: surgical sterilization, double barrier method of contraception, local contraception;

Exclusion Criteria:

* Refusal to participate;
* Hypersensitivity to propofol, dexmedetomidine;
* Prolonged mechanical ventilation in case of surgical complications (bleeding, inadequate perfusion of the myocardium);
* Occurred ischemic stroke;
* History of the ischemic stroke;
* History of the neurodegenerative diseases;
* History of the mental disorders;
* Use of neuroleptics, antidepressants for the last 5 years;
* History of the cardiac surgery in the past;
* Patients with chronic pulmonary disease (GOLD 3-4)
* Patients with asthma (moderate or severe),
* Participation in any other clinical trial;
* Gastric or duodenal ulcer with risk of bleeding;
* Chronic renal failure (ClCr less than 50 ml / h)
* Acute renal failure that occurred during surgery (ClCr less than 50 ml / h, or a decrease in the rate of diuresis to 0.1 ml / h in the first 4 hours after surgery and does not respond to diuretic therapy)
* Chronic hepatic insufficiency if there are laboratory signs of hypo coagulation without the use of anticoagulant therapy (INR> 1.5)
* If the patient has not stopped taking anticoagulants or antiplatelet agents in the preoperative period: warfarin 5 days before surgery, clopidogrel 5-7 days before surgery, xarelto / pradaxa 3 days before surgery),
* History of the hematological disease;
* Alcohol abuse in the anamnesis (3-4 times a week).
* Condition after chemotherapy;
* Pregnancy, lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
vasopressor requirements | every hour during sedation(up to 12 hours)
  incidence of cases of using norepinephrine. measurement tool is a fact of using that is marked as yes\no in the check-list
dose of norepinephrine | every hour during sedation (up to 12 hours)
  measure the maximum dose of norepinephrine in mcg\kg\min to achieve mean arterial pressure 70 mmHg

SECONDARY OUTCOMES:
Length of stay in the ICU | before discharging from ICU to the ward ( up to 3 days)
  measure at days

CONTACTS AND LOCATIONS:
Overall Officials: Yelyzaveta Plechysta, MD, Principal Investigator — Chief of the anesthesia department
Locations (1):
- Cardiosurgery departments with intensive care block, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No